CLINICAL TRIAL: NCT03948360
Title: A First-In-Human Pilot Study of a Novel Wearable Phototherapy System for the Management of Acute Burn Wounds
Brief Title: Safety Study of a Novel Wearable Phototherapy System for the Management of Acute Burn Wounds
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rogers Sciences Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Device Feasibility
Other Study IDs: BOS1705
Record Dates: First submitted 2018-11-15; First posted 2019-05-13 (Actual); Last update posted 2019-05-13 (Actual); Status verified 2019-05

CONDITIONS: Burn Wound
Keywords: acute burn, thermal injury, wound, phototherapy, wound healing, antimicrobial
MeSH Terms: conditions — Burns; Wounds and Injuries | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: The study model is sequential. Arm I will consist of the first 3 participants, with each participant receiving LIMB phototherapy over standard of care (SOC). The subsequent participants will comprise Arm II, with each participant to receive only LIMB phototherapy without standard of care. Dose modifications of the phototherapy can be made in Arm II, and will be determined based on any treatment-related adverse events observed in Arm I. Up to 12 participants in total will be enrolled.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- LIMB Phototherapy with SOC (Experimental): Arm I: The first 3 participants enrolled will receive standard of care therapy under the Low-Irradiance Monochromatic Biostimulation (LIMB) phototherapy device.
  Interventions: Device: Low-Irradiance Monochromatic Biostimulation (LIMB) Device; Other: Standard of Care
- LIMB Phototherapy without SOC (Experimental): Arm II: The subsequent participants will receive only the Low-Irradiance Monochromatic Biostimulation (LIMB) phototherapy device without standard of care.
  Interventions: Device: Low-Irradiance Monochromatic Biostimulation (LIMB) Device

INTERVENTIONS:
Device: Low-Irradiance Monochromatic Biostimulation (LIMB) Device — The LIMB System is a portable and wearable phototherapeutic system that consists of a Light Patch and Power Pack. The Power Pack delivers power to the Light Patch, which attaches to the participant and emits blue spectrum (405nm low-irradiance) light. The Light Patch contains an array of thin optical arrays that evenly illuminate the surface. The Power Pack is powered by a Lithium Thionyl Chloride (Li-SOCI2) battery.
Other: Standard of Care — Standard of care therapy as defined for this clinical trial is standard gauze dressing soaked in Sulfamylon (mafenide acetate) solution.
  Arms: LIMB Phototherapy with SOC

SUMMARY:
The primary purpose of this first-in-human, early feasibility study is to assess safety and feasibility of the Low-Irradiance Monochromatic Biostimulation (LIMB) System as a phototherapeutic intervention for the management of acute burn wounds. The prototype LIMB device will be evaluated for the occurrence of adverse events (treatment-related or otherwise) of the LIMB System, a portable, wearable, light-emitting system developed by Rogers Sciences, Inc. (RSI). The device will be administered in the small feasibility pilot to confirm design, usability and operating specifications that will inform procedures and endpoints of a subsequent large, multicenter clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving care at Shriners Hospitals for Children-Boston for a skin tissue injury.
* Patients who have at least one wound with exposed area sufficient, in the Investigator's opinion, to receive LIMB therapy.
* Willing and able to adhere to daily LIMB therapy protocol.

Exclusion Criteria:

* Patients deemed not medically stable by the treating Investigator.
* Patients with clinical signs and symptoms of systemic infection at baseline.
* Patients with burn wounds limited to their head and genitalia.
* Patients who, in the opinion of the Investigator, will not require daily dressing changes.
* Patients receiving photosensitizing agents that result in cutaneous phototoxicity prior to enrollment. Patients who have received one or more of the following photosensitizers cannot be enrolled into the study: photofrin, amiodarone, chloropromazine, fluoroquinolone antibiotics, thiazide diuretics, quinine, demethylchlortetracycline, psoralens, nalidixic acid, tetracycline, naproxen.
* Patients currently enrolled or participating in another investigational device, drug or biological trial within 30 days of the Screening Visit.
* Patients currently receiving any bandages or devices containing silver compounds.
* Patients on a ventilator, who have fluid resuscitation or are in any terminal condition.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Estimated)
Dates: Start 2017-09-07 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Occurrence of Adverse Events from LIMB Phototherapy as Assessed by CTCAE v4.0 | up to 7 days
  To evaluate the occurrence of adverse events (treatment-related or otherwise) from LIMB phototherapy from the time of device application up to 7 days. Reporting consistent with CTCAE v4.0. Duration of LIMB phototherapy can be shortened per discretion of treating Investigator.

SECONDARY OUTCOMES:
Change in Bioburden assessed through Wound Culture | up to 7 days
  To evaluate the effect of LIMB phototherapy on microbial bioburden. Wound culture specimens are collected at each daily dressing change to measure the change in microbial bioburden when compared to baseline.

OTHER OUTCOMES:
Change in Pain as Assessed by Checklist Pain Behavior Scale | up to 7 days
  To evaluate the change in participant's pain score during LIMB phototherapy treatment. Pain assessments taken daily at dressing change.

CONTACTS AND LOCATIONS:
Overall Officials: Robert L. Sheridan, MD, Principal Investigator — Shriners Hospitals for Children-Boston
Locations (1):
- Shriners Hospitals for Children-Boston, Boston, Massachusetts, United States